CLINICAL TRIAL: NCT04274036
Title: Evaluation of Stigma and Related Factors in Fibromyalgia Patients
Brief Title: Evaluation of Stigma and Related Factors in Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif GÜLER, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: 13
Record Dates: First submitted 2020-02-13; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Social Support; Stigma
MeSH Terms: conditions — Fibromyalgia; Social Stigma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia Patients: Fibromyalgia patients diagnosed according to the 2016 American College of Rheumatology criteria.
- Healthy-Controls: Healthy controls without pain or chronic illness

SUMMARY:
Stigmatization is especially studied in mental disorders such as schizophrenia. In recent years, different chronic diseases such as AIDS, tuberculosis, and diabetes have also been shown to decrease in quality of life due to the "stigma" of these patients.

DETAILED DESCRIPTION:
Stigmatization is especially studied in mental disorders such as schizophrenia. In recent years, different chronic diseases such as AIDS, tuberculosis, and diabetes have also been shown to decrease in quality of life due to the "stigma" of these patients. Fibromyalgia patients with chronic widespread body pain and accompanying subjective fatigue, depression, and anxiety; Although there is no objective pathology from the outside, it can be stigmatized in family life, work-life and health institutions they apply for the diagnosis of pain due to the intensive complaints. The fact that the subjective complaints seen without an objective pathology are so severe makes the management of these patients difficult. To reveal the presence of stigma in patients diagnosed with fibromyalgia compared with the healthy control group is the main aim of this study. It is the secondary purpose of this study to determine related factors such as gender, age, educational status, marital status, employment status, income level, pain duration, pain intensity, medications used, and social support received from patients' family and the environment. We hypothesize that this group of patients suffers more stigma and the quality of life decreases due to this stigma.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* To be diagnosed with fibromyalgia according to American College of Rheumatology 2016 revised criteria

Exclusion Criteria:

* Have been diagnosed and treated with fibromyalgia before
* Presence of any diagnosis that can cause secondary fibromyalgia (rheumatic diseases such as rheumatoid arthritis, ankylosing spondylitis)
* The presence of anemia
* Vitamin D deficiency
* Presence of known endocrine, neurological and cardiac diseases
* Antidepressant use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fibromiyalgia patients and healthy controls with an allocation ratio of 2:1.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline
  A scale to measure pain which "0" shows no pain and "10" shows worst pain ever
Discomfort Intolerance Scale | Baseline
  The Discomfort Intolerance Scale is brief, self-report index of the degree to which individuals tolerate physical discomfort including pain. Items for this scale were developed by experts in pain and anxiety. Participants rate the questions on a scale ranging from 0 (not at all like me) to 6 (extremely like me). Higher points show worst outcomes.
The Distress Tolerance Scale | Baseline
  Distress tolerance is defined as the capacity to experience and withstand negative psychological states. Distress may be the result of cognitive or physical processes but manifests in an emotional state often characterized by action tendencies to alleviate the emotional experience. Distress tolerance is considered a meta-emotion construct that consists of one's evaluations and expectations of experiencing negative emotional states in respect to tolerability and aversiveness, appraisal and acceptability, tendency to absorb attention and disrupt functioning, and regulation of emotions, specifically, the consequent strength of action tendencies to either avoid or immediately attenuate the experience
Fibromyalgia Impact Questionnaire - Revised | Baseline
  The revised Fibromyalgia Impact Questionnaire has 21 individual questions All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'.
Stigma Scale for Chronic Illness | Baseline
  The stigma scale consists of 24 items. Item scores range from 1 (never) to 5 (always). A summary index is calculated by adding all scores, ranging from 24 to 120, with higher scores reflecting the worst stigmatization.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Taksim Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No